CLINICAL TRIAL: NCT03091205
Title: Proper Extent of Maze Intercaval Lesion
Acronym: Maze
Status: Withdrawn | Type: Observational
Why Stopped: Unable to obtain funding source
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 017-048
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It's hypothesized that a mean and range distance from the cavo-atrial junction to the area where there is complete loss of conductive tissue can be measured to better inform surgeons performing the Cox-Maze procedure. A patient scheduled for any cardiac surgery where visualization and mapping of cavo-atrial junction is possible could be entered into the study if they meet the inclusion/exclusion requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years male or female
* Scheduled for any cardiac surgery where visualization and mapping of cavo-atrial junction is possible
* Subjects willing and able to provide written informed consent

Exclusion Criteria:

* Subjects receiving surgery with non-sternotomy access
* Presence of or history of transvenous pacing leads
* Subjects receiving a re-do cardiac surgery
* Subjects with a history of pericarditis
* Subjects who are in atrial fibrillation or atrial flutter and cannot be converted out of it.
* Any medical condition or finding for which the Investigator used medical discretion to determine the subject should be excluded
* Subject is currently participating in another clinical trial.
* Subject is unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for any cardiac surgery where visualization and mapping of cavo-atrial junction is possible
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-04-15 (Estimated)

PRIMARY OUTCOMES:
Distance until complete loss of conductive tissue | 6 Months
  To measure the mean and range distance from the cavo-atrial junction to the area where there is complete loss of conductive tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy George, M.D, Principal Investigator — Baylor Reasearch Institute
Locations (1):
- The Heart Hospital Baylor Plano, Plano, Texas, United States